CLINICAL TRIAL: NCT00421668
Title: A Trial of Zinc and Micronutrients in Tanzanian Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christopher Duggan, Professor of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD048969
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diarrheal Illnesses; Respiratory Illness; Growth Faltering
Keywords: HIV; Tanzania; Micronutrients; Infants/children; Infectious Disease; Growth faltering
MeSH Terms: conditions — Communicable Diseases | interventions — Zinc; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Multivitamins (Experimental): Vitamins C, E, B1, B2, niacin, B6, folate, and B12
  Interventions: Drug: Multivitamins
- Multivitamins + Zinc (Experimental): Vitamins C, E, B1, B2, niacin, B6, folate and B12, and zinc
  Interventions: Drug: Zinc; Drug: Multivitamins
- Zinc (Experimental): zinc
  Interventions: Drug: Zinc
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc — zinc
  Arms: Multivitamins + Zinc; Zinc
Drug: Multivitamins — Vitamins C, E, B1, B2, niacin, B6, folate and B12
  Arms: Multivitamins; Multivitamins + Zinc
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized clinical trial of multiple micronutrients, zinc, zinc + micronutrients, or placebo among 2400 children born to HIV-negative Tanzanian mothers.

DETAILED DESCRIPTION:
We propose to study the efficacy of zinc or multiple micronutrient supplementation in reducing the risk of infectious diseases and growth faltering among infants and young children in Tanzania. Infants born to HIV-negative women will be recruited and randomly assigned in a factorial design to either zinc, micronutrients (vitamins C, E, B1, B2, niacin, B6, folate and B12), micronutrients plus zinc, or a placebo given daily. Children will be followed at monthly clinic visits from age 6 weeks for 18 months. Data obtained will include socioeconomic status, anthropometric data (weight, length, head circumference, and arm anthropometrics), dietary intake (including breastfeeding duration and frequency), hemoglobin, ferritin, and blood smear for malaria. The primary outcomes will be the incidence of diarrhea and respiratory tract infections. Secondary outcomes will be weight and length gain. A subset of children will be tested for blood concentrations of vitamin A, E, zinc and C-reactive protein. All children will receive a large periodic dose of vitamin A every 6 months as per standard of care in Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, live born infants born to HIV- negative women
* Mothers will need to have registered for pre-natal care before 34 weeks gestation
* intend to stay in Dar es Salaam for until delivery and 18 months thereafter.

Exclusion Criteria:

* infants born with multiple congenital abnormalities

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | from ages 6 weeks to 18 months
respiratory tract infections | from ages 6 weeks to 18 months

SECONDARY OUTCOMES:
Weight gain | from age 6 weeks to 18 months
Length/height gain | from age 6 weeks to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Duggan, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimbili Uinverstiy College of Health Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Liu E, Manji KP, Kirby MA, Kisenge R, Lauer JM, Fawzi WW, Sudfeld CR, Duggan CP. Effects of Zinc Supplementation on Metabolomic Profiles in Tanzanian Infants: A Randomized Trial. J Nutr. 2024 Feb;154(2):403-411. doi: 10.1016/j.tjnut.2023.12.011. Epub 2023 Dec 11. PMID 38092153
- [Derived] Rees CA, Kisenge R, Manji KP, Liu E, Fawzi WW, Duggan CP. Identifying Infants and Young Children at Risk of Unplanned Hospital Admissions and Clinic Visits in Dar es Salaam, Tanzania. Pediatr Infect Dis J. 2020 Dec;39(12):e428-e434. doi: 10.1097/INF.0000000000002875. PMID 32842043
- [Derived] Lauer JM, McDonald CM, Kisenge R, Aboud S, Fawzi WW, Liu E, Tran HQ, Gewirtz AT, Manji KP, Duggan CP. Markers of Systemic Inflammation and Environmental Enteric Dysfunction Are Not Reduced by Zinc or Multivitamins in Tanzanian Infants: A Randomized, Placebo-Controlled Trial. J Pediatr. 2019 Jul;210:34-40.e1. doi: 10.1016/j.jpeds.2019.02.016. Epub 2019 Apr 2. PMID 30952509
- [Derived] Blakstad MM, Smith ER, Etheredge A, Locks LM, McDonald CM, Kupka R, Kisenge R, Aboud S, Bellinger D, Sudfeld CR, Fawzi WW, Manji K, Duggan CP. Nutritional, Socioeconomic, and Delivery Characteristics Are Associated with Neurodevelopment in Tanzanian Children. J Pediatr. 2019 Apr;207:71-79.e8. doi: 10.1016/j.jpeds.2018.10.066. Epub 2018 Dec 14. PMID 30559023
- [Derived] Etheredge AJ, Manji K, Kellogg M, Tran H, Liu E, McDonald CM, Kisenge R, Aboud S, Fawzi W, Bellinger D, Gewirtz AT, Duggan CP. Markers of Environmental Enteric Dysfunction Are Associated With Neurodevelopmental Outcomes in Tanzanian Children. J Pediatr Gastroenterol Nutr. 2018 Jun;66(6):953-959. doi: 10.1097/MPG.0000000000001978. PMID 29613921
- [Derived] Winje BA, Kvestad I, Krishnamachari S, Manji K, Taneja S, Bellinger DC, Bhandari N, Bisht S, Darling AM, Duggan CP, Fawzi W, Hysing M, Kumar T, Kurpad AV, Sudfeld CR, Svensen E, Thomas S, Strand TA. Does early vitamin B12 supplementation improve neurodevelopment and cognitive function in childhood and into school age: a study protocol for extended follow-ups from randomised controlled trials in India and Tanzania. BMJ Open. 2018 Feb 22;8(2):e018962. doi: 10.1136/bmjopen-2017-018962. PMID 29472265
- [Derived] Locks LM, Mwiru RS, Mtisi E, Manji KP, McDonald CM, Liu E, Kupka R, Kisenge R, Aboud S, Gosselin K, Gillman M, Gewirtz AT, Fawzi WW, Duggan CP. Infant Nutritional Status and Markers of Environmental Enteric Dysfunction are Associated with Midchildhood Anthropometry and Blood Pressure in Tanzania. J Pediatr. 2017 Aug;187:225-233.e1. doi: 10.1016/j.jpeds.2017.04.005. Epub 2017 May 9. PMID 28499715
- [Derived] Locks LM, Manji KP, Kupka R, Liu E, Kisenge R, McDonald CM, Aboud S, Wang M, Fawzi WW, Duggan CP. High Burden of Morbidity and Mortality but Not Growth Failure in Infants Exposed to but Uninfected with Human Immunodeficiency Virus in Tanzania. J Pediatr. 2017 Jan;180:191-199.e2. doi: 10.1016/j.jpeds.2016.09.040. Epub 2016 Nov 7. PMID 27829511
- [Derived] Locks LM, Manji KP, McDonald CM, Kupka R, Kisenge R, Aboud S, Wang M, Bellinger DC, Fawzi WW, Duggan CP. The effect of daily zinc and/or multivitamin supplements on early childhood development in Tanzania: results from a randomized controlled trial. Matern Child Nutr. 2017 Apr;13(2):e12306. doi: 10.1111/mcn.12306. Epub 2016 May 18. PMID 27189038
- [Derived] McDonald CM, Manji KP, Gosselin K, Tran H, Liu E, Kisenge R, Aboud S, Fawzi WW, Gewirtz AT, Duggan CP. Elevations in serum anti-flagellin and anti-LPS Igs are related to growth faltering in young Tanzanian children. Am J Clin Nutr. 2016 Jun;103(6):1548-54. doi: 10.3945/ajcn.116.131409. Epub 2016 Apr 27. PMID 27121948
- [Derived] Locks LM, Manji KP, McDonald CM, Kupka R, Kisenge R, Aboud S, Wang M, Fawzi WW, Duggan CP. Effect of zinc and multivitamin supplementation on the growth of Tanzanian children aged 6-84 wk: a randomized, placebo-controlled, double-blind trial. Am J Clin Nutr. 2016 Mar;103(3):910-8. doi: 10.3945/ajcn.115.120055. Epub 2016 Jan 27. PMID 26817503
- [Derived] McDonald CM, Manji KP, Kisenge R, Aboud S, Spiegelman D, Fawzi WW, Duggan CP. Daily Zinc but Not Multivitamin Supplementation Reduces Diarrhea and Upper Respiratory Infections in Tanzanian Infants: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Nutr. 2015 Sep;145(9):2153-60. doi: 10.3945/jn.115.212308. Epub 2015 Jul 22. PMID 26203094